CLINICAL TRIAL: NCT02758847
Title: Evaluation of Paclitaxel in Patients With CLI (Critical Limb Ischemia) and Femoropopliteal Occlusive Disease Treated With DCB Angioplasty
Brief Title: Evaluation of Paclitaxel in Patients With CLI and Femoropopliteal Occlusive Disease Treated With DCB Angioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabih A. Chaer (Other)
Responsible Party: Sponsor-Investigator, Rabih A. Chaer, Professor of Surgery, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO15120093
Record Dates: First submitted 2016-04-11; First posted 2016-05-03 (Estimated); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Ischemia
Keywords: critical lower limb ischemia with tissue loss
MeSH Terms: conditions — Ischemia | interventions — Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Critical Limb Ischemia (CLI) and Tissue Loss (Other): Paclitaxel® coated balloons will be used for patients identified with Critical Limb Ischemia (CLI) and Tissue Loss. Patients with CLI will receive either Angiogram, Medtronic DCB (paclitaxel)/stent or Angiogram, Bard DCB (paclitaxel)/stent
  Interventions: Device: Angiogram, Medtronic DCB (paclitaxel)/stent; Device: Angiogram, Bard DCB (paclitaxel)/stent

INTERVENTIONS:
Device: Angiogram, Medtronic DCB (paclitaxel)/stent — Paclitaxel® coated balloons will be used for patients identified with Critical Limb Ischemia (CLI) and Tissue Loss. Each participant will receive angiogram with DCB (drug coated balloon)/stenting with wound debridement. 50% of subjects will receive an Angiogram, Medtronic DCB (paclitaxel)/stent. Tissue samples will be sent to pathology for specific staining to evaluate trace evidence of the drug paclitaxel.
Device: Angiogram, Bard DCB (paclitaxel)/stent — Paclitaxel® coated balloons will be used for patients identified with Critical Limb Ischemia (CLI) and Tissue Loss. 50% of subjects will receive 'Angiogram, Bard DCB (paclitaxel)/stent' . Tissue samples will be sent to pathology for specific staining to evaluate trace evidence of the drug paclitaxel.

SUMMARY:
The use of drug coated balloon (DCB) in patients with critical limb ischemia (CLI) and tissue loss has recently raised some concerns after the IN.PACT deep trial using paclitaxel coated balloon angioplasty in the tibial arteries was terminated. The investigators objective is to establish the safety and efficacy of drug coated balloon (DCB) for femoropopliteal occlusive disease in patients with critical limb ischemia (CLI) and tissue loss.

The investigators objective is to establish the safety and efficacy of drug coated balloon (DCB) for femoropopliteal occlusive disease in patients with critical limb ischemia (CLI) and tissue loss.

DETAILED DESCRIPTION:
Although the association between the drug coated balloon (DCB) therapy and limb outcomes could not be clearly linked to the use of antiproliferative agents, the findings of paclitaxel crystals downstream of the treated lesions, although in small amounts, has raised concerns about the safety of such therapy in patients with critical limb ischemia (CLI) and tissue loss.

These concerns, however, may not translate to patients with femoropopliteal occlusive disease as the amount of paclitaxel reaching the foot may be even smaller after being filtered by the calf musculature.

Since the use of DCB angioplasty in the Superficial Femoral Artery (SFA) and popliteal has been shown to deliver significantly more durable outcomes compared to standard angioplasty alone, with reported primary patency rates of almost 90% at one year, this therapy may even be more needed in patients with tissue loss where prolonged patency is essential for wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Patient population: all patients with CLI (critical limb ischemia) and tissue loss scheduled for endovascular intervention for femoral popliteal occlusive or multilevel disease.
* Patient or patient's legal representative have been informed of the nature of the study, agrees to participate and has signed an Ethical Committee approved consent form
* Female patients of childbearing potential have a negative pregnancy test ≤7 days before the procedure and are willing to use a reliable method of birth control for the duration of study participation
* Patient has documented chronic Critical Limb Ischemia (CLI) in the target limb prior to the study procedure with Rutherford Category 5 or 6
* General Angiographic Inclusion Criteria
* Single or multiple lesions with ≥70% diameter stenosis (DS) of different lengths in the SFA and/or popliteal arteries.
* Iliac inflow or Tibial outflow interventions can be done at the discretion of the investigator with standard balloon Percutaneous Transluminal Angioplasty (PTA)

Exclusion Criteria:

* Patient unwilling or unlikely to comply with Follow-Up schedule
* Aneurysm in the target vessel
* Acute thrombus in the target limb
* Sensitivity to Paclitaxel
* Immunosuppressed patients (transplant, chemotherapy, etc.)

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rabih A Chaer, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Judith Brimmeier, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
still early in the recruitment process

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Critical Limb Ischemia (CLI) and Tissue Loss
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Critical Limb Ischemia (CLI) and Tissue Loss
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Diabetes [Count of Participants; unit: Participants] | 38

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing
Description: Percentage of participants with wound healing defined as > 50% area/volume reduction of baseline ulcer(s) in the treated leg at 1 year.
Time Frame: 12 months
Population: 50 consecutive patients with documented Rutherford Category 5 or 6 chronic limb threatening ischemia (CLTI) in the target limb were prospectively enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Critical Limb Ischemia (CLI) and Tissue Loss
Number analyzed (Participants) | 50
Participants | 30

2. Primary Outcome: Amputation Free Survival
Description: Percentage of participants with a 6 month amputation free survival.
Time Frame: 6 months
Population: The study patients that are alive and have follow up information at 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Critical Limb Ischemia (CLI) and Tissue Loss
Number analyzed (Participants) | 35
percentage of participants | 71.4

3. Secondary Outcome: Primary Patency ( Determine if Vessel Remains Open)
Description: Prospective duplex ultrasound will be performed at the listed interval to verify (primary and secondary) patency of targeted vessels. Primary patency is defined as the target vessel "patency obtained without the need for additional or secondary surgical or endovascular procedures (the interval from the time of the original intervention until any intervention designed to maintain or re-establish patency is performed)."
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Critical Limb Ischemia (CLI) and Tissue Loss
Number analyzed (Participants) | 50
percentage of participants | 97

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a 1 year period
Description: The definition of adverse events does not differ from the clinical trials.gov Definitions
Arm/Group | Critical Limb Ischemia (CLI) and Tissue Loss
All-Cause Mortality (participants affected / at risk) | 16/50
Serious Adverse Events (participants affected / at risk) | 11/50
Other Adverse Events (participants affected / at risk) | 12/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Critical Limb Ischemia (CLI) and Tissue Loss (N=50)
Major Amputation (Vascular disorders) | 11 (11) — Major Limb Amputations is defined as either a below the knee or above the knee amputation of the lower extremity
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Critical Limb Ischemia (CLI) and Tissue Loss (N=50)
Wound Infection (Infections and infestations) | 12 (12) — Wound Infections are defined as clinical scenarios that necessitate treatment with antibiotics for a diagnosis of a wound infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT02758847/Prot_SAP_000.pdf